CLINICAL TRIAL: NCT01299025
Title: Balance Training for People With Multiple Sclerosis Using Nintendo Wii Fit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro County Council (Other Government)
Collaborators: Uppsala-Örebro Regional Research Council (Other); Norrbacka-Eugenia Foundation (Other)
Responsible Party: Principal Investigator, Anette Forsberg, PhD, PhD, Research physical therapist, Örebro County Council
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ö28-10
Record Dates: First submitted 2011-02-17; First posted 2011-02-18 (Estimated); Results first posted 2015-04-24 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Multiple Sclerosis
Keywords: balance; walking
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Participants allocated as controls receive no treatment. They may be physically active as usual.
- Training with Nintendo Wii Fit (Experimental): Training 6 weeks with Nintendo Wii Fit, 30 minutes 2 times per week
  Interventions: Other: Training using Nintendo Wii Fit

INTERVENTIONS:
Other: Training using Nintendo Wii Fit — Training 2 times per week, 30 minutes, for 6 weeks.
  Arms: Training with Nintendo Wii Fit

SUMMARY:
The aim is to evaluate balance training using Nintendo Wii Fit. The hypothesis is that a period of training will increase balance capacity och self-efficacy.

People with diagnosed multiple sclerosis are invited to participate. Estimation of study power gave that 29 people in each group was necessary to detect a difference in the primary outcome measure, Timed Up and Go test.

Other measures used are the Four square step test, Dynamic Gait Index, Timed stands test, 25 foot walking test, 12-item Walking scale and the ABC scale.

Participants were randomised to either training or control. The training consisted of 6 weeks training with Nintendo Wii Fit 30 minutes 2 times a week.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed multiple sclerosis
* Subjective experience of affected balance and walking
* Being able to walk 100 meters with assistance

Exclusion Criteria:

* Cognitive or language deficits that prevents using the self-rating scales
* Visual deficits that prevents training with television games
* Weight above 149 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anette Forsberg, PhD, Principal Investigator — Örebro County Council
Locations (4):
- Sweden (4):
  - Mälarsjukhuset, Eskilstuna
  - Karlstad hospital, Karlstad
  - Family Medicine Research centre, Örebro
  - Västerås hospital, Västerås

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Training With Nintendo Wii Fit
Started | 42 | 42
Completed | 39 | 41
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Training With Nintendo Wii Fit | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (11.1) | 50.0 (11.5) | 49.8 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 64
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  Sweden | 42 | 42 | 84

OUTCOME MEASURES:

1. Primary Outcome: Change in Timed Up and Go Test From Day 1 to Day 42
Description: Change in seconds on the Timed Up and Go test (TUG). In the TUG test time is taken from rising from a chair, walking 3 meters, turning,walking back and sitting down.
Time Frame: Measured at day 1 (before the training period) and at day 42 (after the training period)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Control | Training With Nintendo Wii Fit
Number analyzed (Participants) | 39 | 41
seconds | 0.1 (2.1) | -0.8 (2.4)
Statistical Analysis 1: Comparison: Control vs Training With Nintendo Wii Fit; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Score on the Dynamic Gait Index From Day 1 to Day 42
Description: The Dynamic Gait index consists of 8 items. Performance on each item is rated from 0 (severe impairment) to 3 (nomal performance). Minimum total score is 0 and maximum 24. Higher scores indicate better walking and balance performance.
Time Frame: Measured at day 1 (before training) and day 42 (after training)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Control | Training With Nintendo Wii Fit
Number analyzed (Participants) | 39 | 41
Scores on a scale | 1.0 (2.0) | 1.78 (2.3)

3. Secondary Outcome: Change in the Activities-specific Balance Confidence (ABC) Scalefrom Day 1 to Day 42
Description: The ABC scale is a self-rating scale of balance activities in everyday Life. It includes 16 items. The patient rates his/her performance from 0-100. Score on each item are summed an divided by 16. Minimum score is 0 and maximum score 100. A higher score indicate higher confidence in ones balance and walking capacity.
Time Frame: Measured at day 1 (before training) and day 42 (after training)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Control | Training With Nintendo Wii Fit
Number analyzed (Participants) | 39 | 41
Scores on a scale | 2.7 (11.8) | 5.0 (14.4)

4. Secondary Outcome: Change in the 12 Item Walking Scale From Day 1 to Day 42
Description: The 12 item walking scale is a self-rating scale of walking limitations. The scale includes 12 items that each are scores from 1 to 5, where 5 is extremely limited. Scores are added and transformed to a scale from 0-100. 0 indicates no limitation and 100 extremely limited.
Time Frame: Measured at day 1 and day 42, before and after the training
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Control | Training With Nintendo Wii Fit
Number analyzed (Participants) | 39 | 41
Scores on a scale | -3.95 (18.1) | -5.9 (11.5)

ADVERSE EVENTS:
Arm/Group | Control | Training With Nintendo Wii Fit
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No